CLINICAL TRIAL: NCT05717491
Title: Study of Diabetes' Risk Factors and Accelerated Aging According to Socio-economic Status in a Population From the North of France
Acronym: PREVENDIAB
Status: Completed | Type: Observational
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: National Center for Precision Diabetic Medicine,PreciDIAB (Unknown)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Medical director of CPSL, Institut Pasteur de Lille
Other Study IDs: 2021-A01727-34
Record Dates: First submitted 2021-12-14; First posted 2023-02-08 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes; PreDiabetes
Keywords: (Pre) diabetes; Risk factors; Precarious; Accelerated aging
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Glucose Intolerance | interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA methylation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main group: Cross-sectional study
  Interventions: Other: Biological analysis, Physical examination and Questionnaires
- Sub group: Case control study
  Interventions: Other: Physical examination and Questionnaires

INTERVENTIONS:
Other: Biological analysis, Physical examination and Questionnaires — Biological analysis, Physical examination and questionnaires will be performed for all patients of the main group.
  Groups: Main group
Other: Physical examination and Questionnaires — In addition to exams for the main group, there will be 2 additional examinations (bone densitometry and arterial stiffness) for the patients of the subgroup and others questionnaires.
  Groups: Sub group

SUMMARY:
Populations in precarious situations or with low socio-economic status have an increased risk of diabetes and accelerated aging. According to the population studied, the elements that can explain these health inequalities are not unequivocal and remain poorly known.

The north of France, particularly affected by socio-economic disparities, has a prevalence of diabetes among the highest in metropolitan France. This is why investigators want to study the clinical, biological, social and behavioural risk factors of the entry into diabetes and accelerated aging among a large population in the North of France.

This study aims to characterize the population (among which a majority (55%) suffers from precarious conditions) who come to carry out their health examination at the Pasteur Institute in Lille in order to study the risk factors to better explain these health inequalities.

This research consists of a main descriptive observational, cross-sectional study carried out on 2233 volunteers (main group) over 18 months, and a complementary analytical case-control study that will be offered to 216 participants (sub-group).

DETAILED DESCRIPTION:
Primary Objective : Assessment of Prevalence of Prediabetes and Diabetes by Socio-Economic Status

Primary efficacy endpoint : Fasting glucose value based on EPICES score :

Glycemia:

* Normal: fasting glucose ≤ 1g/l
* Prediabetes: fasting glucose >1 g/l and ≤1.25 g/l
* Diabetes: fasting glucose >1.25 g/l

EPICES score: quintiles of score distribution (Q1 to Q5)

Secondary Objectives specific to the main group:

* Characterize the population and analyze the risk factors (clinical, biological, socio-economic and behavioural) of diabetes and prediabetes in this population.
* Study the level of biological ageing and factors associated with accelerated ageing.
* Estimate the risk of (pre)diabetes and accelerated aging based on socio-economic profile.

Secondary Objectives specific to the sub-group:

* Assess the impact of economic, social and cultural capital on health in terms of diabetes and accelerated aging.
* Analyze the effect on diabetes and accelerated aging of the exposures assessed: body composition, physical activity, arterial rigidity, cognitive status, psychiatric disorders, fragility, pain.

Secondary endpoints specific to the main group: :

* Prevalence ratio of diabetes and prediabetes calculated for:

  * Clinical, paraclinical parameters (Oral examination, Muscle strength,Advanced glycation products) and anthropometric parameters (medical history, height, weight, BMI, Waist and hip circumference, Neck circumference, body composition measurement, Systolic and diastolic blood pressure, Unipedal stance test).
  * Biological (blood and genetic).
  * Behavioural/environmental predictors: (socio-economic status, physical activity(RICCI GAGNON), diet(HDI), quality of life (MQLI), stress-anxiety(PSS), toxic habits, fragility(FRIED) ).
* Assessment of the level of ageing

  * Biological Aging Marker: DNAmPhenoAge (DNA methylation phenotypic age)
  * Accelerated ageing: age regression DNAmPhenoAge on chronological age
  * Analysis of age-related parameters (inflammatory, renal, hormonal, body composition measurement, fragility, advanced glycation products, muscle strength) and correlation with methylation rate and DNAmPhenoAge.
* Prevalence ratio of (pre)diabetes and accelerated aging according to socio-economic status

  * Evaluation of (pre)diabetes: fasting blood sugar
  * Accelerated Aging Assessment: DNAm PhenoAge
  * Social Status Assessment: EPICES Q1 to Q5 Score
  * Assessment of economic status: Income level

Secondary endpoints specific to the subgroup:

* Risk (OR) of (pre)diabetes and accelerated aging according to social, economic, cultural and marital status

  * Evaluation of (pre)diabetes: fasting blood sugar
  * Accelerated Aging Assessment: DNAmPhenoAge
  * Socio-economic and cultural criteria

    * Social status (EPICES score)
    * Economic status (income)
    * Cultural status (semi-directive interview)
    * Professional status (educational level, socio-professional category, marital status)
* Risk (OR) of (pre)diabetes and accelerated aging for assessed exposures:

  * Evaluation of (pre)diabetes: fasting blood sugar
  * Accelerated Aging Assessment: DNAmPhenoAge
  * Exposure Assessment

    * Arterial Stiffness Index
    * Body composition (mineral density, lean mass, fat mass) (DEXA test)
    * Insomnia Severity Index (ISI)
    * Cognitive Status (MOCA)
    * Physical Activity (GPAQ Questionnaire)
    * Alcohol consumption (FACE)
    * Psychiatric disorders (MINI)
    * Fragility (REFS score)
    * Pain Scale (EVA)

ELIGIBILITY:
Inclusion Criteria:

* Adult, male or female
* Consultant for the health prevention examination at the Examination Centre of Health of the Institut Pasteur of Lille
* Available to follow the constraints generated by the study
* Signature of the informed consent
* Status of insured person in France

Exclusion Criteria:

* Participation in another clinical study or in a period of exclusion from another study
* Adult deprived of liberty or under judicial protection
* Impediment to give the free and informed consent (understanding, persons under guardianship/curators, etc.)
* Incompatible scheduling
* Other reason (state of health or concomitant treatments,...) considered by the principal investigator or a qualified co-investigator not compatible with the proper conduct of the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Populations in precarious situations or with a low socioeconomic level have an increased risk of entering diabetes and aging accelerated. Depending on the populations studied, the elements that could explain these health inequalities are not unequivocal and are still badly known.
  The Hauts-de-France region, particularly affected by disparities socio-economic, has one of the most prevalent diabetes high in the metropolis. This is why it's important to study the factors clinical, biological, social and behavioral risks of entry in diabetes and accelerated aging in a large population of North of France.
  This study aims to characterize the population of the Centre's consultants of Health Examinations at the Institut Pasteur de Lille, of which a majority (55%) suffers from precarious conditions, in order to study the risk factors to better explain these health inequalities.
Sampling Method: Non-Probability Sample
Enrollment: 2014 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Fasting glucose value according to the level of precariousness | Day 0
  Glycemia in g/L Level of precariousness given by EPICES score

SECONDARY OUTCOMES:
Prevalence ratio of (pre)diabetes calculated for clinical, biological and behavioral/environmental explanatory variables | Day 0
  In %
Assessment of the level of accelerated ageing (DNAmPhenoAge) | Day 0
  In units of years
Prevalence ratio of (pre) diabetes and accelerated aging according to the socio-economic status | Day 0
  In %
Risk (odds Ratio) of (pre) diabetes and accelerated aging according to social, economic, cultural and professional status | Until Day 90
  Without units
Risk (odds Ratio) of (pre) diabetes and accelerated aging for assessed exposures | Until Day 90
  Without units

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Dr FROGUEL, PhD, Study Chair — PRECIDIAB; Matthias Mr VANDESQUILLE, PhD, Study Director — PRECIDIAB
Locations (1):
- Institut Pasteur de Lille, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Center for Precision Medicine on Diabetes - PreciDIAB — https://www.precidiab.org/en/precidiab-national-center-for-precision-medicine-on-diabetes/